CLINICAL TRIAL: NCT03368807
Title: An Objective Assessment of Mealtime Bolus Insulin Behavior and Associated Factors
Brief Title: Assessment of Mealtime Bolus Insulin Behavior
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 16866; F3Z-MC-IOQV (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-11-30; First posted 2017-12-11 (Actual); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring; Insulin Lispro

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Blinded CGM (Continuous Glucose Monitoring): Participants received Insulin lispro 100 U/mL (units per millilitre) injected via the pen and they were blinded to CGM device recording as directed in study period 1.
  Interventions: Device: Continuous Glucose Monitoring; Drug: Insulin Lispro
- Unblinded CGM: Participants received Insulin lispro 100 U/mL injected via the pen and they were unblinded to CGM device recording as directed in study period 2.
  Interventions: Device: Continuous Glucose Monitoring; Drug: Insulin Lispro

INTERVENTIONS:
Device: Continuous Glucose Monitoring — Commercially available
Drug: Insulin Lispro — As prescribed.

SUMMARY:
The main purpose of this study is to estimate missed bolus insulin doses in diabetics. This is a 12-week, single-arm, outpatient, exploratory study with two study periods in Type 1 or Type 2 diabetics, with an investigational reusable injection pen, insulin, and a Continuous Glucose Monitoring (CGM) device.

ELIGIBILITY:
Inclusion Criteria:

* Have a Type 1 Diabetes Mellitus (T1D) or a Type 2 Diabetes Mellitus (T2D) diagnosis
* Must be taking a mealtime bolus dose insulin, greater than or equal to (≥) 3 doses
* Each individual bolus insulin dose must be less than (<) 40 units
* Must be taking a stable insulin dose regimen for the last 3 months
* Must be taking a bolus insulin analog (for example insulin lispro [U-100]/[U-200], insulin aspart, or insulin glulisine). In addition, must be able to switch to insulin lispro U-100 for the duration of the trial
* Must have a hemoglobin A1c (HbA1c) ≥8.0% in the last 6 months
* Participants with T1D must be ≥21 to less than or equal to (≤) 65 years of age. Participants with T2D must be ≥35 to ≤65 years of age
* Women of childbearing potential must meet the following: (Note: females of childbearing potential are defined as those who have experienced menarche and who are NOT permanently sterile or postmenopausal. Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause)

  * Must agree to use 1 highly effective method of contraception, or a combination of 2 effective methods of contraception for the entirety of the study
  * Must test negative for pregnancy as indicated by a negative serum or urine pregnancy test
* Participants with prior CGM/flash glucose monitoring experience must have stopped CGM/flash glucose monitoring ≥3 months prior to enrollment

Exclusion Criteria:

* Have known tape/adhesive allergies with CGM sensors
* Medical conditions, visual, physical, psychiatric, or cognitive impairment(s) that may preclude the ability to participate in the trial
* Have history of liver disease, acute or chronic hepatitis, or alanine aminotransferase or aspartate aminotransferase levels ≥3 times the upper limit of the reference range within the last 6 months
* Have history of chronic kidney disease stage 4 and higher within the last 6 months, or history of renal transplantation
* Have active malignancy
* Are pregnant or planning to become pregnant
* Are on or are intending to begin a weight loss program
* Participants with T1D who have taken off-label antihyperglycemic agents within last 3 months
* Have received insulin by continuous subcutaneous insulin infusion in the last 3 months
* Participants taking opioid medications for medically invalid reasons or at doses considered excessive
* Participants on routine use of acetaminophen
* Currently undergoing systemic treatment with:

  * Immunosuppressive medication
  * Chronic (lasting longer than 2 weeks) systemic glucocorticoid therapy (excluding topical and inhaled preparations) or have received such therapy within the prior 2 weeks
* Are currently enrolled in any other clinical study involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study
* Have participated, within the last 30 days, in a clinical study involving an investigational product
* Are unwilling or unable to comply with the use of a data collection device to directly record data

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 1 and Type 2 Diabetics
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (6):
  - AMCR Institute, Inc., Escondido, California
  - Science 37 Inc, Los Angeles, California
  - Coastal Metabolic Research Ctr, Ventura, California
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Iowa Diabetes & Endocrinology Research Center, West Des Moines, Iowa
  - Advanced Research Institute, Ogden, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wolpert H, Rodbard D, Xue J, Johnson J, Dassau E. Characterizing insulin dosing behaviour and glycaemic excursions: Development of metrics using connected insulin pen and continuous glucose monitoring. Diabetes Obes Metab. 2025 May;27(5):2507-2514. doi: 10.1111/dom.16249. Epub 2025 Feb 10. PMID 39930566

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Period 1/Study Period 2: Participants with type 1 diabetes or type 2 diabetes received prescribed insulin regimen suitable for their disease state using insulin lispro 100 units per millilitre (U/mL) injected via the pen. During the study, participants had their glucose monitored via the continuous glucose monitoring (CGM) device, which was blinded during Study Period 1 and unblinded during Study Period 2.
Period: Period 1 (Blinded CGM)
Arm/Group | Study Period 1/Study Period 2
Started | 79
Received at Least 1 Dose of Study Drug | 78
Completed | 73
Not Completed | 6
Not completed — Withdrawal by Subject | 3
Not completed — Protocol Violation | 1
Not completed — Sponsor Decision | 1
Not completed — Lost to Follow-up | 1
Period: Period 2 (Unblinded CGM)
Arm/Group | Study Period 1/Study Period 2
Started | 73
Completed | 73
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received study drug.
Groups:
- Overall Study: Participants received prescribed insulin regimen suitable for their disease state using insulin lispro 100 U/mL injected via the pen. During the study, participants had their glucose monitored via the CGM device, which was blinded during Study Period 1 and unblinded during Study Period 2.
Arm/Group | Overall Study
Number analyzed (Participants) | 79
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.01 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 66
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 73
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 79
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 30.9 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Days Per Month With a Missed Bolus Insulin Dose With Blinded CGM
Description: The average number of days per month with a missed bolus insulin dose was calculated in participants with Type 1 Diabetes or Type 2 Diabetes using blinded CGM measurements and the pen. The time of insulin dosing and glucose excursions were assessed using the display times recorded by the pen and CGM devices, respectively.
Time Frame: Week 1 up to 6 weeks
Population: All enrolled participants who received at least one dose of study drug and have missed bolus insulin dose data.
Measure: Mean (Standard Deviation); unit: Days per month
Groups:
- Blinded CGM: Participants received Insulin lispro 100 U/mL injected via the pen and they were blinded to CGM device recording as directed.
Arm/Group | Blinded CGM
Number analyzed (Participants) | 68
Days per month | 19.3 (6.2)

2. Secondary Outcome: Average Number of Days Per Month With a Missed Bolus Insulin Dose With Unblinded CGM
Description: The average number of days per month with a missed bolus insulin dose was calculated in participants with Type 1 Diabetes or Type 2 Diabetes using unblinded CGM measurements and the pen. The time of insulin dosing and glucose excursions were assessed using the display times recorded by the pen and CGM devices, respectively
Time Frame: Week 6 up to 12 weeks
Population: All enrolled participants who received at least one dose of study drug and have missed bolus insulin dose data.
Measure: Mean (Standard Deviation); unit: Days per month
Groups:
- Unblinded CGM: Participants received Insulin lispro 100 U/mL injected via the pen and they were unblinded to CGM device recording as directed.
Arm/Group | Unblinded CGM
Number analyzed (Participants) | 65
Days per month | 17.9 (5.7)

3. Secondary Outcome: Percentage of Time-in-Range (Glucose >70 and ≤180 Milligrams Per Deciliter) With Blinded CGM
Description: Percentage of time-in-range (glucose >70 and ≤180 milligrams per deciliter) was calculated in participants with Type 1 Diabetes or Type 2 Diabetes based on blinded CGM data collected in the study period. The time component of the time-in-range statistic was calculated using the display time recorded by the CGM device.
Time Frame: Baseline up to 6 weeks
Population: All enrolled participants who received at least one dose of study drug and have data for Percentage of Time-in-Range.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Blinded CGM
Number analyzed (Participants) | 68
Percentage of time | 42.7 (18.8)

4. Secondary Outcome: Percentage of Time-in-Range (Glucose >70 and ≤180 Milligrams Per Deciliter) With Unblinded CGM
Description: Percentage of time-in-range (glucose >70 and ≤180 milligrams per deciliter) was calculated in participants with Type 1 Diabetes or Type 2 Diabetes based on unblinded CGM data collected in the study period. The time component of the time-in-range statistic was calculated using the display time recorded by the CGM device.
Time Frame: Week 6 up to 12 weeks
Population: All enrolled participants who received at least one dose of study drug and have data for Percentage of Time-in-Range.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Unblinded CGM
Number analyzed (Participants) | 65
Percentage of time | 49.6 (20.0)

5. Secondary Outcome: Percentage of Missed Bolus Doses Per Month With Blinded CGM
Description: Percentage of missed bolus doses per month was estimated in participants with Type 1 diabetes or Type 2 diabetes using blinded CGM measurements and the pen.
Time Frame: Baseline up to 6 weeks
Population: All enrolled participants who received at least one dose of study drug and have data for missed bolus doses.
Measure: Mean (Standard Deviation); unit: Percentage of missed bolus dose
Arm/Group | Blinded CGM
Number analyzed (Participants) | 68
Percentage of missed bolus dose | 25.3 (12.3)

6. Secondary Outcome: Percentage of Missed Bolus Doses Per Month With Unblinded CGM
Description: Percentage of missed bolus doses per month was estimated in participants with Type 1 diabetes or Type 2 diabetes using unblinded CGM measurements and the pen.
Time Frame: Week 6 up to 12 weeks
Population: All enrolled participants who received at least one dose of study drug and have data for missed bolus doses.
Measure: Mean (Standard Deviation); unit: Percentage of missed bolus dose
Arm/Group | Unblinded CGM
Number analyzed (Participants) | 65
Percentage of missed bolus dose | 23.3 (10.2)

7. Secondary Outcome: Average Number of Missed Bolus Insulin Doses Per Day With Blinded CGM
Description: The average number of missed bolus doses per day was estimated in participants with Type 1 diabetes or Type 2 diabetes using blinded CGM measurements and the pen.
Time Frame: Baseline up to 6 weeks
Population: All enrolled participants who received at least one dose of study drug and have data for missed bolus doses.
Measure: Mean (Standard Deviation); unit: Dose per day
Arm/Group | Blinded CGM
Number analyzed (Participants) | 68
Dose per day | 0.9 (0.4)

8. Secondary Outcome: Average Number of Missed Bolus Insulin Doses Per Day With Unblinded CGM
Description: The average number of missed bolus doses per day was estimated in participants with Type 1 diabetes or Type 2 diabetes using unblinded CGM data.
Time Frame: Week 6 up to 12 weeks
Population: All enrolled participants who received at least one dose of study drug and have data for missed bolus doses.
Measure: Mean (Standard Deviation); unit: Dose per day
Arm/Group | Unblinded CGM
Number analyzed (Participants) | 65
Dose per day | 0.9 (0.4)

9. Secondary Outcome: Average Number of Missed and Suboptimal Bolus Dose (MSBD) Events Per Month With Blinded CGM
Description: The number of Missed and Suboptimal Doses (MSBDs) per month was calculated in participants with Type 1 Diabetes or Type 2 Diabetes as the sum of the identified missed bolus doses and suboptimal bolus doses for each participant for each period.
Time Frame: Baseline up to 6 weeks
Population: All enrolled participants who received at least one dose of study drug and have data for missed bolus doses.
Measure: Mean (Standard Deviation); unit: Dose per month
Arm/Group | Blinded CGM
Number analyzed (Participants) | 68
Dose per month | 68.3 (24.1)

10. Secondary Outcome: Average Number of Missed and Suboptimal Bolus Dose (MSBD) Events Per Month With Unblinded CGM
Description: as for outcome 9
Time Frame: Week 6 up to 12 weeks
Population: All enrolled participants who received at least one dose of study drug and have data for missed bolus doses.
Measure: Mean (Standard Deviation); unit: Dose per month
Arm/Group | Unblinded CGM
Number analyzed (Participants) | 65
Dose per month | 61.9 (22.2)

ADVERSE EVENTS:
Time Frame: Up To 12 Weeks
Description: All enrolled participants who received at least one dose of study drug.
Arm/Group | Blinded CGM | Unblinded CGM
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/73
Serious Adverse Events (participants affected / at risk) | 3/78 | 2/73
Other Adverse Events (participants affected / at risk) | 22/78 | 9/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinded CGM (N=78) | Unblinded CGM (N=73)
Chest pain (General disorders) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Medical device removal (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinded CGM (N=78) | Unblinded CGM (N=73)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Application site bruise (General disorders) | 1 (1) | 0 (0)
Application site pain (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Device damage (Product Issues) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diabetic microangiopathy (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Some investigators wait until a multi-site publication is published (or 2 years if not published sooner) plus a 90 day review period.

DOCUMENTS (2):
  • Study Protocol (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT03368807/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT03368807/SAP_001.pdf